# Hualien Tzu Chi Hospital Medical TechnologyResearch Project Proposal In the hospital

| A. Basic II | niormatio | П | Application | on number · | |
|---|---|---|---|---|---|
| | | | Project: The principal in | nvestigator of this | project is a |
| | senior member of our institution. | | | | |
| Project Category<br>(Single choice) | Experimental Research (up to 800,000 NT Dollars) Non-experimental Research (up to 400,000 NT Dollars) | | | | |
| | | | ` • ′ | , | 000 NT D - 11 ) |
| | | - | artment Project (Maxim | • | JOU NT Dollars) |
| | , | - | ment Heads for Applica<br>Project (Up to 200,000 | | |
| | | | aboration Research Pro | | 00 NT Dollars) |
| | | - | roject of the Ministry of | | , |
| | | | 800,000 NT Dollars) | Science and Tech | illology |
| | | | Lesearch Project (Up to | 400 000 NT Doll: | ars) |
| 人員類別 | | aucutton 1 | toscuron rioject (op to | 100,000 1(1 2011 | w15) |
| (單選) | Physician | | □Non-Physicia | | |
| The Project | | - | igmatic breathing in p | | _ |
| Name | interaction: impact on gastrointestinal and psychological symptoms as well a<br>autonomic nervous system | | | | |
| Principal | autonomic ne | ervous sysi | em | Applicant | |
| Investigator | Wong, | Job Title | Attending Physician | Department or | Gastroenterology |
| Name | Ming-Wun | 300 11110 | rttenamg i mysician | Division | Gustroenterology |
| Project | Project | | | | |
| Execution | From Septem | ber 1, 202 | 23 to December 31, 202 | 4, a total of 1 year | r. |
| Deadline | | | | | |
| | | | ch Applied Research | h <u>l</u> Techno | ological |
| | Development | | and in annlied was an | ah and taahnala | deal development |
| Nature and | | | aged in applied resear<br>gory of innovative rese | | |
| Classification of | | | ch & Development Clas | | |
| Research | | | earch $\square(3)$ Medical | | |
| | | | dical Assistance Opera | | |
| | | 。 | arear rissistance open | | er, preuse speerry |
| H 1: 4: C | Holistic Care | Classifica | ntion: | | |
| Holistic Care (Please refer to | (1) Patient- | | ( physiological | psychological | environmental |
| the noun | spiritual) | | ( <b>—</b> F ) = | <b>—</b> F=9===8== | |
| explanations, | (2) Health Ed | lucation ( | behavior change | ge∏health pr | omotion Disease |
| multiple | Prevention | ` | | , <u> </u> | _ |
| selections | | , , | Treatment) | | |
| allowed) | (3) Other, ple | | , | | 0 |
| Has the current in | n-house projec | t ever app | lied for the 112th-year | Ministry of Scien | ce and Technology |
| Special Research | Project? | No TY | es | | |
| | Has any application been made for government grants for various research projects in the current | | | | |
| year? | Yes, Total | <u>1</u> items | | | |
| - | | | of 1 research project v | within the institut | e. (Projects co-led |
| with others will n | | / | | | |
| The priority orde | The priority order of this project is <u>1</u> . | | | | |

| 2 | | | | | | |
|---|---|---|---|---|---|---|
| Does this project | require No H | uman | experiments/human | specimens | (including | human |
| embryos/human er | nbryonic stem cells) | Animal | l Experimentation | | | |
| ☐Biosafety (inclu | ding recombinant DNA | exper | iments/genetically me | odified field | trials/secon | ıd-level |
| or higher infectiou | s biological materials) ' | ? <b>[</b> Ple | ase check | | | |
| 3 | Name: <u>Wong, Ming-W</u><br>E-MAIL: <u>hypertr42@g</u> | | • , , | 825#13224 | / 0982-0988 | 12 |

**B.** Apply for Financial Assistance (Budget allocation will be included in the review scoring criteria; please do not inflate the budget.)

In accordance with the actual needs of the research project, subsidies can be applied for the following items: For individual research projects, the upper limit for experimental researchers is 800,000 NT dollars, and for non-experimental researchers, the principle upper limit is 400,000 NT dollars. For newly recruited personnel research projects, the total research budget is capped at 200,000 NT dollars. For university-industry collaborative research projects, the total research budget is capped at 400,000 NT dollars. For projects under the Department of Whole Person Care, the budget ceiling is 800,000 NT dollars. Technology transfer projects within the Ministry of Science and Technology have a maximum budget limit of 800,000 NT dollars.

| Subsidy Programs | | Requested Amount |
|---|---|---|
| | 1. Research personnel expenses | 83,016 |
| Business expenses | 2. Animal testing expenses | |
| | 3. Consumables,<br>Supplies, Books, and<br>Miscellaneous expenses | 716,984 |
| Research equipment expenses | | |
| | Total | 800,000 |

# **C.** Equipment configuration

The principal instruments required for this project, their respective locations, and the signatures of the individuals authorized to use them. •

| Instrument Name | Location Setup (Department) | Signature of the Unit<br>Supervisor/Manager agreeing |
|---|---|---|
| | | to the use of the equipment |

# D. Personnel involved in the project

1. Mainly researching human resources

| Category (Host, co-host, co-presenter, research assistant, etc.) | Name | Current position | Nature, projects, and scope of work involved in this research project. |
|---|---|---|---|
| Host | Wong, Ming-<br>Wun | Attending Physician of Gastroenterology | Project schedule supervision, research progress tracking and plan development, data analysis and report writing. |
| Co-host | Chen, Chien-<br>Lin | Director of Gastroenterology | Actual case handling procedures, such as inspection operations, in the planned project. |
| Co-host | Yi, Chih-Hsun | | Actual case handling procedures, such as inspection operations, in the planned project. |
| Co-host | Liu, Tso-Tsai | Director of Endoscopy Department | Actual case handling procedures, such as inspection operations, in the planned project. |
| Co-host | Lei, Wei-Yi | Attending Physician of Gastroenterology | Actual case handling procedures, such as inspection operations, in the planned project. |
| Co-host | Hung, Jui-<br>Sheng | Attending Physician of Gastroenterology | Actual case handling procedures, such as inspection operations, in the planned project. |
| Research assistant | Chen, Yan-Zhu | | Organize data, data analysis and statistics and handle administrative affairs. |
| Research assistant | Jian,Yu-xuan | | Organize data, data analysis and statistics and handle administrative affairs. |

2. Research projects that the host, co-hosts, and co-researchers have participated in in the past three years.

| | past tince years. | | 1 | |
|---|---|---|---|---|
| Surname name | Count painting name say | Jobs within the plan | From year to month | Grant agencies |
| Wong,<br>Ming-Wun | Antireflux mucosal ablation for the treatment of PPI-dependent gastroesophageal reflux disease: treatment efficacy and physiological alteration | Host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong, | Exploring pathophysiological mechanisms of laryngopharyngeal reflux: utilization with artificial intelligence and clinical implication for precision diagnosis and personalized treatment strategies | Host | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology |
| Wong,<br>Ming-Wun | Supervised Learning Artificial Intelligence in 24-<br>h Impedance-pH: Technique Performance and<br>Clinical Implications for Diagnosing GERD | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong,<br>Ming-Wun | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden in patients with disorders of long COVID gut brain interaction a doub le blind, randomized,placebo controlled study | Co-host | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |
| | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong, | Relevance of esophageal hypervigilance, functional gastrointestinal disorders, and psychological distress as pathophysiological | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |

| vei | rsion date: (Version 4,11/13/2023) | | 1 | |
|---|---|---|---|---|
| | mechanisms to esophageal symptoms | | | |
| Wong,<br>Ming-Wun | Oropharyngeal swallowing physiology in patients with esophageal hypomotility: Studies with HRPM | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong,<br>Ming-Wun | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic implications for esophageal dysfunction and gastroesophageal reflux disease | Co-host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |
| Wong,<br>Ming-Wun | Utility of high resolution pharyngeal manometry and Sydney Swallow Questionnaire for evaluation of oropharyngeal dysphagia and voice disorder | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong, | Application of Artificial Intelligence in High-<br>resolution Esophageal Function Testing: A Study<br>on Unsupervised Deep Learning Algorithms | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong, | Impact of regulating diet and exercise on clinical characteristics and intestinal microbiota in patients with metabolic-related fatty liver | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong,<br>Ming-Wun | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Wong,<br>Ming-Wun | Diagnosis and establishment of indications for<br>proton pump inhibitors in the improvement of<br>laryngopharyngeal reflux based on nighttime<br>average basal impedance values of the proximal<br>esophagus | Host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Wong,<br>Ming-Wun | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | Co-host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Wong,<br>Ming-Wun | Exploring the role of esophageal microbiome in<br>the novel impedance parameters, clinical<br>classification, and hypersensitivity in<br>gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong,<br>Ming-Wun | Exploring the interrelationship and pathogenesis of esophageal acid sensitivity, esophageal secondary peristalsis, and subtypes of gastroesophageal reflux | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Wong,<br>Ming-Wun | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug<br>response | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Chen,<br>Chien-Lin | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden in patients with disorders of long COVID gut brain interaction a doub le blind, randomized,placebo controlled study | Host | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Chen,<br>Chien-Lin | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | Host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Chen, | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic | Host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |

| Vei | rsion date: (Version 4,11/13/2023) | | | |
|---|---|---|---|---|
| | implications for esophageal dysfunction and | | | |
| | gastroesophageal reflux disease | | | |
| Chan | Jing Si Herbal Tea in the treatment of dyspeptic | | 2022/1/1 | Tzu Chi |
| Chen, | symptoms and psychophysical burden | Host | 2022/1/1~ | Medical |
| Chien-Lin | by improving and pay anophysical caraci | 11000 | 2022/12/31 | Corporation |
| | | | | Corporation |
| | Exploration of esophageal reflux clearance, | | | |
| Chen, | mucosa integrity, and psychological | | 2022/1/1~ | Hualien Tzu |
| | characteristics: pathophysiological and | Host | 2022/12/31 | Chi Hospital |
| Chien-Lin | therapeutic implications for gastroesophageal | | 2022/12/31 | Cili Hospitai |
| | reflux disease | | | |
| | Relevance of esophageal hypervigilance, | | | |
| Chen, | functional gastrointestinal disorders, and | _ | 2023/01/01~ | Hualien Tzu |
| | psychological distress as pathophysiological | Co-host | 2023/12/31 | Chi Hospital |
| Chien-Lin | 1 1 2 | | 2023/12/31 | Cili Hospitai |
| | mechanisms to esophageal symptoms | | | |
| Chen, | Antireflux mucosal ablation for the treatment of | | 2023/01/01~ | Hualien Tzu |
| | PPI-dependent gastroesophageal reflux disease: | Co-host | 2023/12/31 | Chi Hospital |
| Chien-Lin | treatment efficacy and physiological alteration | | 2023/12/31 | Cili Hospitai |
| Chen, | Oropharyngeal swallowing physiology in patients | | 2022/01/01 | H1: T |
| Chen, | with esophageal hypomotility: Studies with | Co-host | 2023/01/01~ | Hualien Tzu |
| Chien-Lin | HRPM | | 2023/12/31 | Chi Hospital |
| | Exploring pathophysiological mechanisms of | | | |
| | | | | Ministry of |
| Chen, | | G 1 . | 2022/8/1~ | Ministry of |
| C1 : I : | artificial intelligence and clinical implication for | | 2025/07/31 | Science and |
| Chien-Lin | precision diagnosis and personalized treatment | | 2020/07/51 | Technology |
| | strategies | | | |
| | Relationships among mucosal afferent | | | |
| CI | innervation, esophageal peristalsis and | | 20 2 2 10 11 | Ministry of |
| Chen, | pharmacological modulation in the human | Co-host | 20 2 2/8/1~ | Science and |
| Chien-Lin | esophagus: implications for pathophysiology and | eo nost | 2025/07/31 | Technology |
| | management in patients with GERD | | | reciniology |
| C1 | Impact of opioids on esophageal peristalsis and | | 2022/1/1 | 11 1: T |
| Chen, | acid reflux characteristics:relevance for | Co-host | 2022/1/1~ | Hualien Tzu |
| Chien-Lin | esophageal pathophysiology and therapeutic | e a nest | 2022/12/31 | Chi Hospital |
| | implications | | | |
| Chen, | Supervised Learning Artificial Intelligence in 24- | | 2022/1/1 | II1: T |
| Chen, | h Impedance-pH: Technique Performance and | Co-host | 2022/1/1~ | Hualien Tzu |
| Chien-Lin | Clinical Implications for Diagnosing GERD | | 2022/12/31 | Chi Hospital |
| | Utility of high resolution pharyngeal manometry | | | |
| Chen, | | Ca hast | 2022/1/1~ | Hualien Tzu |
| Chion Lin | and Sydney Swallow Questionnaire for evaluation | Co-host | 2022/12/31 | Chi Hospital |
| Cinen-Lin | of oropharyngeal dysphagia and voice disorder | | | 1 |
| Chen, | Application of Artificial Intelligence in High- | | 2022/1/1~ | Hualien Tzu |
| | resolution Esophageal Function Testing: A Study | Co-host | 2022/17/1 | Chi Hospital |
| Chien-Lin | on Unsupervised Deep Learning Algorithms | | 2022/12/31 | Cili Hospitai |
| | Impact of regulating diet and exercise on clinical | | 0000/1/1 | II 1: T |
| Chen, | characteristics and intestinal microbiota in | Co-host | 2022/1/1~ | Hualien Tzu |
| Chien-Lin | patients with metabolic-related fatty liver | | 2022/12/31 | Chi Hospital |
| | Exploring the role of esophageal microbiome in | | | |
| Chen, | 1 0 | | 2021/1/1 | Huglian Tax |
| Chell, | the novel impedance parameters, clinical | Host | 2021/1/1~ | Hualien Tzu |
| Chien-Lin | classification, and hypersensitivity in | | 2021/12/31 | Chi Hospital |
| | gastroesophageal reflux disease | | | |
| | Exploring the interrelationship and pathogenesis | | | |
| Chen, | of esophageal acid sensitivity, esophageal | C - 1 | 2021/1/1~ | Hualien Tzu |
| Chian Lin | secondary peristalsis, and subtypes of | Co-host | 2021/12/31 | Chi Hospital |
| Chien-Lin | gastroesophageal reflux | | | Γ |
| I | 10 | | | |


| 70 | rsion date • (Version 4,11/13/2023) | | | |
|---|---|---|---|---|
| Chen,<br>Chien-Lin | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug<br>response | | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Chen,<br>Chien-Lin | Relationships among mucosal afferent innervation, esophageal peristalsis and pharmacological modulation in the human esophagus: implications for pathophysiology and management in patients with GERD | Co-host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Chen,<br>Chien-Lin | Diagnosis and establishment of indications for<br>proton pump inhibitors in the improvement of<br>laryngopharyngeal reflux based on nighttime<br>average basal impedance values of the proximal<br>esophagus | Co-host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Chen,<br>Chien-Lin | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | Host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Yi, Chih-<br>Hsun | Jing Si Herbal Tea in the treatment of dyspeptic<br>symptoms and psychophysical burden in patients<br>with disorders of long COVID gut brain<br>interaction a doub le blind, randomized,placebo<br>controlled study | Co-host | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Yi, Chih-<br>Hsun | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Relevance of esophageal hypervigilance, functional gastrointestinal disorders, and psychological distress as pathophysiological mechanisms to esophageal symptoms | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Antireflux mucosal ablation for the treatment of PPI-dependent gastroesophageal reflux disease: treatment efficacy and physiological alteration | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Oropharyngeal swallowing physiology in patients with esophageal hypomotility: Studies with HRPM | | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic implications for esophageal dysfunction and gastroesophageal reflux disease | Co-host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |
| Yi, Chih-<br>Hsun | Exploration of esophageal reflux clearance, mucosa integrity, and psychological characteristics: pathophysiological and therapeutic implications for gastroesophageal reflux disease | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Impact of opioids on esophageal peristalsis and acid reflux characteristics:relevance for esophageal pathophysiology and therapeutic implications | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Utility of high resolution pharyngeal manometry and Sydney Swallow Questionnaire for evaluation of oropharyngeal dysphagia and voice disorder | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |

| Ve | rsion date: (Version 4,11/13/2023) | | | |
|---|---|---|---|---|
| Yi, Chih-<br>Hsun | Application of Artificial Intelligence in High-<br>resolution Esophageal Function Testing: A Study<br>on Unsupervised Deep Learning Algorithms | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Supervised Learning Artificial Intelligence in 24-h Impedance-pH: Technique Performance and Clinical Implications for Diagnosing GERD | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Impact of regulating diet and exercise on clinical characteristics and intestinal microbiota in patients with metabolic-related fatty liver | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Yi, Chih-<br>Hsun | Exploring the interrelationship and pathogenesis of esophageal acid sensitivity, esophageal secondary peristalsis, and subtypes of gastroesophageal reflux | Host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Exploring the role of esophageal microbiome in<br>the novel impedance parameters, clinical<br>classification, and hypersensitivity in<br>gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug<br>response | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Yi, Chih-<br>Hsun | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Yi, Chih-<br>Hsun | Impact of regulating diet and exercise on clinical characteristics and intestinal microbiota in patients with metabolic-related fatty liver | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Jing Si Herbal Tea in the treatment of dyspeptic<br>symptoms and psychophysical burden in patients<br>with disorders of long COVID gut brain<br>interaction a doub le blind, randomized,placebo<br>controlled study | Co-host | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Liu, Tso-<br>Tsai | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Relevance of esophageal hypervigilance, functional gastrointestinal disorders, and psychological distress as pathophysiological mechanisms to esophageal symptoms | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Oropharyngeal swallowing physiology in patients with esophageal hypomotility: Studies with HRPM | | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Antireflux mucosal ablation for the treatment of PPI-dependent gastroesophageal reflux disease: treatment efficacy and physiological alteration | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic implications for esophageal dysfunction and gastroesophageal reflux disease | Co-host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |


| ve | rsion date: (Version 4,11/13/2023) | | | |
|---|---|---|---|---|
| Liu, Tso-<br>Tsai | Exploration of esophageal reflux clearance, mucosa integrity, and psychological characteristics: pathophysiological and therapeutic implications for gastroesophageal reflux disease | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Impact of opioids on esophageal peristalsis and acid reflux characteristics:relevance for esophageal pathophysiology and therapeutic implications | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Utility of high resolution pharyngeal manometry<br>and Sydney Swallow Questionnaire for evaluation<br>of oropharyngeal dysphagia and voice disorder | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Supervised Learning Artificial Intelligence in 24-<br>h Impedance-pH: Technique Performance and<br>Clinical Implications for Diagnosing GERD | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Application of Artificial Intelligence in High-<br>resolution Esophageal Function Testing: A Study<br>on Unsupervised Deep Learning Algorithms | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Liu, Tso-<br>Tsai | Exploring the role of esophageal microbiome in<br>the novel impedance parameters, clinical<br>classification, and hypersensitivity in<br>gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Exploring the interrelationship and pathogenesis of esophageal acid sensitivity, esophageal secondary peristalsis, and subtypes of gastroesophageal reflux | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug<br>response | Co host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Liu, Tso-<br>Tsai | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | Co-host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Lei, Wei-<br>Yi | Relevance of esophageal hypervigilance, functional gastrointestinal disorders, and psychological distress as pathophysiological mechanisms to esophageal symptoms | Host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Relationships among mucosal afferent innervation, esophageal peristalsis and pharmacological modulation in the human esophagus: implications for pathophysiology and management in patients with GERD | Host | 2022/8/1~<br>2025/07/31 | Ministry of<br>Science and<br>Technology |
| Lei, Wei-<br>Yi | Impact of opioids on esophageal peristalsis and acid reflux characteristics:relevance for esophageal pathophysiology and therapeutic implications | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden in patients with disorders of long COVID gut brain interaction a doub le blind, randomized,placebo | Co-host | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |


| 1 | rsion date : (Version 4,11/13/2023) | | <u> </u> | |
|---|---|---|---|---|
| | controlled study | | | |
| Lei, Wei-<br>Yi | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Oropharyngeal swallowing physiology in patients with esophageal hypomotility: Studies with HRPM | | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Antireflux mucosal ablation for the treatment of PPI-dependent gastroesophageal reflux disease: treatment efficacy and physiological alteration | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic implications for esophageal dysfunction and gastroesophageal reflux disease | Co-host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |
| Lei, Wei-<br>Yi | Exploration of esophageal reflux clearance, mucosa integrity, and psychological characteristics: pathophysiological and therapeutic implications for gastroesophageal reflux disease | | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Utility of high resolution pharyngeal manometry<br>and Sydney Swallow Questionnaire for evaluation<br>of oropharyngeal dysphagia and voice disorder | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Application of Artificial Intelligence in High-<br>resolution Esophageal Function Testing: A Study<br>on Unsupervised Deep Learning Algorithms | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Supervised Learning Artificial Intelligence in 24-<br>h Impedance-pH: Technique Performance and<br>Clinical Implications for Diagnosing GERD | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Impact of regulating diet and exercise on clinical characteristics and intestinal microbiota in patients with metabolic-related fatty liver | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Lei, Wei-<br>Yi | Relationships among mucosal afferent innervation, esophageal peristalsis and pharmacological modulation in the human esophagus: implications for pathophysiology and management in patients with GERD | Host | 2020/8/1~<br>2022/07/31 | Ministry of<br>Science and<br>Technology |
| Lei, Wei-<br>Yi | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |
| Lei, Wei-<br>Yi | Exploring the role of esophageal microbiome in the novel impedance parameters, clinical classification, and hypersensitivity in gastroesophageal reflux disease | | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Lei, Wei-<br>Yi | Exploring the interrelationship and pathogenesis of esophageal acid sensitivity, esophageal secondary peristalsis, and subtypes of gastroesophageal reflux | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |

| 10. | rsion date: (Version 4,11/13/2023) | | | |
|---|---|---|---|---|
| Lei, Wei-<br>Yi | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug<br>response | | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Oropharyngeal swallowing physiology in patients with esophageal hypomotility: Studies with HRPM | Host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Utility of high resolution pharyngeal manometry<br>and Sydney Swallow Questionnaire for evaluation<br>of oropharyngeal dysphagia and voice disorder | Host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden in patients with disorders of long COVID gut brain interaction a doub le blind, randomized,placebo controlled study | | 2023/01/01~<br>2023/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Hung, Jui-<br>Sheng | Interaction among supragastric belching, psychologic distress and esophageal acid reflux: Implications for optimal management of GERD | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Relevance of esophageal hypervigilance, functional gastrointestinal disorders, and psychological distress as pathophysiological mechanisms to esophageal symptoms | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Antireflux mucosal ablation for the treatment of PPI-dependent gastroesophageal reflux disease: treatment efficacy and physiological alteration | Co-host | 2023/01/01~<br>2023/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Exploring capsaicin sensitization, sensorimotor function, psychophyiological reflux characteristics in human esophagus: therapeutic implications for esophageal dysfunction and gastroesophageal reflux disease | Co-host | 2023/8/1~<br>2026/07/31 | Ministry of<br>Science and<br>Technology |
| Hung, Jui-<br>Sheng | Exploration of esophageal reflux clearance, mucosa integrity, and psychological characteristics: pathophysiological and therapeutic implications for gastroesophageal reflux disease | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Impact of opioids on esophageal peristalsis and acid reflux characteristics:relevance for esophageal pathophysiology and therapeutic implications | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Supervised Learning Artificial Intelligence in 24-<br>h Impedance-pH: Technique Performance and<br>Clinical Implications for Diagnosing GERD | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Application of Artificial Intelligence in High-<br>resolution Esophageal Function Testing: A Study<br>on Unsupervised Deep Learning Algorithms | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Impact of regulating diet and exercise on clinical characteristics and intestinal microbiota in patients with metabolic-related fatty liver | Co-host | 2022/1/1~<br>2022/12/31 | Hualien Tzu<br>Chi Hospital |
| Hung, Jui-<br>Sheng | Jing Si Herbal Tea in the treatment of dyspeptic symptoms and psychophysical burden | Co-host | 2022/1/1~<br>2022/12/31 | Tzu Chi<br>Medical<br>Corporation |
| Hung, Jui-<br>Sheng | Clinical application of high-resolution impedance<br>pharyngeal function examination in the study of<br>pharyngeal swallowing difficulties and drug | | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |

| | response | | | |
|---|---|---|---|---|
| C1 | Exploring the role of esophageal microbiome in<br>the novel impedance parameters, clinical<br>classification, and hypersensitivity in<br>gastroesophageal reflux disease | Co-host | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| G1 | Exploring the interrelationship and pathogenesis of esophageal acid sensitivity, esophageal secondary peristalsis, and subtypes of gastroesophageal reflux | | 2021/1/1~<br>2021/12/31 | Hualien Tzu<br>Chi Hospital |
| C1 | Interrelationships among esophageal peristalsis, mucosa integrity, and mucosa afferent innervation: mechanisms for esophageal dysfunction and gastroesophageal reflux | Co-host | 2020/8/1~<br>2023/07/31 | Ministry of<br>Science and<br>Technology |

# E. Research-related expenses

| Project Name | Explanation | Unit price | Quantity | Total<br>Price | Notes |
|---|---|---|---|---|---|
| 1.Research manpower costs (please consult the Human Resources Department for related insurance expenses) | (1) Dedicated Personnel (Limited to Individual Project Applications): Remuneration for work (including year-end bonus) is the responsibility of the employer for labor insurance and health insurance. The employer is also responsible for labor retirement benefits (insured at 6% of salary) (2) "Part-time staff (must be current students): Work remuneration | 4,400<br>936<br>26<br>1,286<br>270 | 12<br>12<br>12<br>12<br>12<br>12 | 52,800<br>11,232<br>312<br>15,432<br>3,240 | Hourly<br>wage<br>\$176<br>25 hours<br>per month.<br>Subtotal:<br>83,016 |
| | | | Subtotal: | 83,016 | NTD |
| 2. Animal testing expenses | | | Subtotal: | | |
| 3. Consumables,<br>Supplies, Books,<br>and<br>Miscellaneous<br>expenses | Participant Allowance Heart rate variability rental | 1,000<br>9,000 | 600<br>12 | 600,000<br>108,000 | |
| | expenses for equipment Computer peripheral consumables expenses: Toner | 5,000 | 1 | 5,000 | |
| | corrisumatores expenses. Toner cartridge, ink cartridge, printer photosensitive drum/photoreceptor, special printing paper, etc. | 3,984 | 1 | 3,984 | |
| | Miscellaneous: Postage and telecommunication expenses, printing expenses, photocopy paper expenses, photocopying expenses, binding expenses, stationery expenses, poster production expenses, computer data | | | | |

| version a | iate : ( version 4,1 | 1/10/2020) | | |
|---|---|---|---|---|
| | | statistical expenses, computer data analysis expenses, thesis submission fees, thesis publication fees, slicing, embedding, and immunostaining expenses | | |
| | | | Subtotal: | 716,984 |
| equipmo<br>(Accordination books, con<br>peripheran not eligib<br>The necessand large-<br>instrumer determined<br>Research | nts will be ed by the Department, and ons for their se will be | | Subtotal: | 0 |
| Total | | | 800,000 | |

# F. Project Abstract

Please provide a brief overview of the key points of this project within 500 words and customize keywords based on the nature of the project.

Patients with disorders of gut-brain interaction (DGBI) often present gastrointestinal symptoms that do not show noticeable irregularities in standard examinations. However, due to unclear causes and a high prevalence rate, this condition often exerts a profound impact on the physical and mental health of patients. The scope of DGBI encompasses conditions such as laryngopharyngeal reflux, functional dyspepsia, and irritable bowel syndrome. Previous research has confirmed that in patients with DGBI, their autonomic nervous system exhibits an imbalance, characterized by decreased parasympathetic activity and dominant sympathetic activity. Diaphragmatic breathing helps reduce the respiratory rate and can stimulate parasympathetic activity while suppressing sympathetic activity. Hence, it is now officially recommended as an effective adjunct therapy for relieving symptoms of gastroesophageal reflux. Accordingly, this study plans to implement a randomized controlled trial, introducing diaphragmatic breathing to patients with DGBI who exhibit normal results in objective examinations. This work allows evaluate changes in their psychophysical symptoms before and after treatment, as well as alterations in the autonomic nervous system.

**Key words**: disorders of gut-brain interaction, psychophysical symptoms, diaphragmatic breathing, autonomic nervous system

#### Background and Objectives of the Research Project G.

Please elaborate on the background, objectives, significance, as well as the domestic and international research status related to this research project. Provide a review of the important references and literature relevant to this project.

# **Research Background**

# Disorders of gut-brain interaction, DGBI

Functional GI Disorders, currently referred to as Disorders of gut-brain interaction (DGBI), encompass gastrointestinal symptoms for which, upon objective examination, no organic cause can be identified. Nevertheless, patients still endure the distressing symptoms related to the gastrointestinal tract. The symptoms of gastrointestinal disorders are diverse, encompassing the esophagus, stomach, small intestine, and large intestine. The origin of these symptoms is complex and includes factors such as imbalance in the intestinal microbiota, changes in mucosal immune function, alterations in signaling around the intestinal area, and dysregulation of central nervous system control over intestinal signaling and motor function (Figure 1).<sup>2</sup> If it affects the upper digestive tract, it may lead to symptoms such as upper abdominal pain and bloating; these symptoms are referred to as Functional Dyspepsia (FD). If it affects the lower digestive tract, there may be issues such as abdominal pain, diarrhea, and constipation; this condition is classified as Irritable Bowel Syndrome (IBS).<sup>2</sup> The recent research we have conducted indicates that among patients with symptoms of gastroesophageal reflux disease (GERD), only about 20% show pathological evidence of reflux. However, among those with throat reflux symptoms (such as hoarseness, sensation of a lump in the throat, chronic cough, and frequent throat clearing), their Esophageal Hypervigilance and Anxiety Scale (EHAS) scores are higher compared to individuals without throat reflux symptoms, even in the absence of pathological reflux evidence.<sup>3</sup> These DGBIs (Functional Gastrointestinal Disorders) do not respond well to conventional gastrointestinal medications, so sometimes it is necessary to supplement treatment with neuromodulators from the field of psychosomatic medicine.<sup>4</sup>

# The Relationship Between the Autonomic Nervous System and the Disorders of gut-brain interaction

The gastrointestinal tract is governed by the intrinsic Enteric nervous system (ENS) and the extrinsic Autonomic nervous system (ANS).5,6 ENS can automatically regulate the gastrointestinal tract, while the Central Nervous System (CNS) interacts with the Enteric Nervous System (ENS) through the Autonomic Nervous System (ANS), providing external neural input to regulate and control gastrointestinal functions (Figure 1).7-9 The Parasympathetic Nervous System (PNS) or Sympathetic Nervous System (SNS), either singly or both, may encounter disruptions, leading to impaired communication between the gastrointestinal tract and the brain, subsequently resulting in Functional Gastrointestinal Disorders (FGID).<sup>5, 10</sup> The upper gastrointestinal tract (esophagus, stomach, small intestine, ascending colon) is innervated by the parasympathetic nervous system, with the main source being the Vagus nerve. In contrast, the lower gastrointestinal tract (transverse colon, descending colon, sigmoid colon, external anal sphincter muscles) receives parasympathetic innervation from the Lumbosacral spinal cord's pre-ganglionic neurons, primarily originating from the S1-S4 segments. 11-13 Most research reports consistently find that patients with Functional Gastrointestinal Disorders (DGBI) exhibit reduced parasympathetic nervous system activity and an increased dominance of sympathetic nervous system activity. These findings align with the autonomic control of gastrointestinal motility: activation of the parasympathetic nervous system enhances E6A0021096-10 Total 30 Page, Page 16

gastrointestinal motility, while activation of the sympathetic nervous system inhibits gastrointestinal motility. 14



**Figure 1**. The possible etiology of DGBI includes microbial imbalance in the intestinal tract, changes in mucosal immune function, alterations in peripheral signaling around the intestines, and dysregulation of central nervous system control over intestinal signaling and motor function. Among these factors, the autonomic nervous system plays a crucial role as a communication bridge between the brain (central) and the gastrointestinal tract (peripheral).<sup>1</sup>

#### Heart rate variability

Early studies have shown that through Heart Rate Variability (HRV), the autonomic nervous system (ANS) can be assessed to evaluate the functional status of the gastrointestinal system. <sup>15, 16</sup> The reason is that the autonomic nervous system (ANS) includes both the parasympathetic and sympathetic nervous systems, which regulate the outgoing and incoming fibers of the gastrointestinal tract through the nucleus tractus solitarius (NTS). The NTS also contains other autonomic neural control over organs whose functions are regulated by the central nervous system (CNS) through the ANS, such as cardiovascular functions. 13, 15 Therefore, the central nervous system (CNS) also influences cardiovascular function through the autonomous regulation of sensory inputs from the gastrointestinal tract. This is because there is interaction between subnuclei in the nucleus tractus solitarius (NTS), regulating the rhythm or variability of the heart, known as heart rate variability (HRV). 13 In addition to assessing the autonomic nervous system (ANS), the analysis of heart rate variability (HRV) has also been found to be clinically effective in evaluating the therapeutic efficacy of the autonomic nervous system for disorders of gut-brain interaction (DGBI). HRV parameters can be used as biological markers for assessing treatment outcomes. 14 For example, electrical stimulation therapy is an emerging treatment method for these diseases.<sup>17</sup> Numerous studies consistently demonstrate that neurostimulation therapy improves symptoms of DGBI by enhancing autonomic nervous system dysfunction assessed through HRV. 18-20

HRV is influenced by two main physiological mechanisms: the first originates from the complex and dynamic interplay between the sympathetic and parasympathetic nervous systems; the second arises from regulatory mechanisms controlling heart rate, including RSA, blood pressure reflexes, and rhythmic variations in vascular tone. HRV is primarily applied in the assessment of the autonomic nervous system (ANS). As follows: 21

#### 1. Time Domain Indicator

- ♦ Root mean square of successive differences (RMSSD): RMSSD reflects the variability between heartbeats and is primarily used to estimate the changes in parasympathetic nervous system activity, especially the vagus nerve, in Heart Rate Variability (HRV).<sup>22</sup> RMSSD is considered to be an important indicator of HRV.<sup>23</sup> The RMSSD values over a 24-hour period are highly correlated with the difference in adjacent normal heartbeat intervals exceeding pNN50 and high-frequency (HF) power.<sup>24</sup> The lower RMSSD values are positively correlated with the risk assessment of sudden unexplained death in epilepsy.<sup>25</sup>
- ♦ Adjacent normal heartbeat interval differences exceeding pNN50: The deviation of adjacent normal heartbeat interval differences beyond pNN50 is closely associated with parasympathetic nervous system activity<sup>26</sup> and is related to RMSSD and HF power. However, RMSSD typically provides a better assessment of parasympathetic nervous system activity (especially in the elderly). Therefore, most researchers tend to choose RMSSD over the adjacent normal-to-normal heartbeat interval differences exceeding pNN50.<sup>27</sup>

#### 2. Frequency Domain Indices

- ♦ Low frequency (LF): The low frequency (LF: 0.04-0.15 Hz) reflects the mixed activity of the sympathetic and parasympathetic nervous systems. In certain situations, LF can be used to assess the influence of the sympathetic nervous system, but this requires consideration of respiratory and other physiological influencing factors.
- ♦ High frequency (HF): The high frequency (HF: 0.15-0.4 Hz) primarily reflects parasympathetic nervous system activity, especially vagal nerve activity. This can be observed through Respiratory Sinus Arrhythmia (RSA).<sup>28</sup>
- ❖ LF/HF ratio : The LF/HF ratio is used to assess the balance between the sympathetic nervous system and the parasympathetic nervous system.

#### Diaphragmatic breathing

The relationship between respiration and the autonomic nervous system (ANS) is closely intertwined, as the phrenic nerve, responsible for controlling the movement of the diaphragm, is connected to the vagus nerve of the parasympathetic nervous system.<sup>29</sup> The respiratory cycle reflects the balance between the parasympathetic and sympathetic nervous systems in the Autonomic Nervous System (ANS), which can be observed through Heart Rate Variability (HRV). The ANS state shifts from the parasympathetic nervous system to the sympathetic nervous system during inhalation, while it transitions from the sympathetic nervous system to the parasympathetic nervous system during exhalation. In HRV, an increase in heart rate indicates enhanced sympathetic nervous system activity during inhalation, whereas a decrease in heart rate signifies increased parasympathetic nervous system activity during exhalation.<sup>30</sup>

Diaphragmatic breathing can be achieved by reducing the respiratory rate, promoting parasympathetic nervous system activity, and concurrently inhibiting sympathetic nervous system activity. <sup>31, 32</sup> Due to the increase in tidal volume during diaphragmatic breathing, the Hering-Breuer reflex is activated. This reflex reduces chemoreflex sensitivity and enhances baroreflex, further lowering sympathetic nervous system activity. <sup>33</sup> The rhythm of diaphragmatic breathing is as follows: Step 1: Inhale through the nose for about 4 seconds, feeling the expansion of the abdomen; Step 2: Hold the breath for 2 seconds; Step 3: Exhale slowly and steadily through the mouth for about 6 seconds (see Figure 2). (Diaphragmatic Breathing for GI Patients - Michigan Medicine) Currently, diaphragmatic breathing is formally recommended for alleviating symptoms of gastroesophageal reflux disease (GERD) and is proven effective in reducing the frequency of reflux occurrences in randomized controlled trials. It is now recognized as an effective adjunctive therapy. <sup>34, 35</sup> However, currently, there is still no randomized controlled experiment confirming the effects of abdominal breathing on other functional gastrointestinal disorders (DGBI issues).



**Figure 2.** Diaphragmatic breathing: When inhaling in the left image, the diaphragm descends, causing the abdomen to protrude. In the right image, during exhalation, the diaphragm ascends, and the abdomen returns to a flat state.

**Figure 3.** During the high-resolution esophageal impedance measurement period after a 20-minute meal, under random allocation, both the healthy control group (a) and the patient group (b) demonstrated a significant reduction in the number of reflux events with diaphragmatic breathing. In contrast, the sham (normal) breathing group showed no significant difference in reflux events.<sup>35</sup>

# **Research Purpose**

For patients with DGBI (Functional Gastrointestinal Disorders) who exhibit gastrointestinal symptoms that cannot identify organic causes after objective examinations, current treatment options are significantly limited. Dysregulation of the autonomic nervous system is one contributing factor. Abdominal breathing, by reducing respiratory frequency, promotes parasympathetic nervous system activity while inhibiting sympathetic nervous system activity. It is now officially recommended by

international consensus conferences as an adjunctive therapy to alleviate symptoms of gastroesophageal reflux.

The purpose of this study is to investigate the autonomic nervous system responses through standardized autonomic nervous system monitoring, focusing on the impact of diaphragmatic breathing on the autonomic nervous system in both healthy subjects and patients with Functional Gastrointestinal Disorders (DGBI). Additionally, the study aims to confirm whether the implementation of diaphragmatic breathing can improve symptoms in DGBI patients, providing a basis for future reference in the treatment of DGBI patients.



# Research hypothesis

#### Hypothesis 1: Diaphragmatic breathing can change Autonomic nervous system

Hypothesis 1-1: Diaphragmatic breathing can increase the activity of the parasympathetic nervous system and decrease the activity of the sympathetic nervous system in healthy subjects.

Hypothesis 1-2: Diaphragmatic breathing can increase parasympathetic nervous system activity and decrease sympathetic nervous system activity in patients with DGBI.

Hypothesis 2: Diaphragmatic breathing can improve symptoms in patients with DGBI.

Hypothesis 2-1: Introducing diaphragmatic breathing can improve symptoms in patients with Laryngopharyngeal Reflux Disease (LPR).

Hypothesis 2-2: Introducing diaphragmatic breathing can improve symptoms in patients with Functional Dyspepsia (FD).

Hypothesis 2-3: Introducing diaphragmatic breathing can improve symptoms in patients with Irritable Bowel Syndrome (IBS).

# H. Research methods, procedures, and execution progress.

- 1.Please elaborate on the research methods adopted in this project and the reasons behind their selection
- 2. Anticipated difficulties and possible solutions.
- 3. If it is a consecutive project, please also attach the annual research progress report or primary data for the corresponding year.

#### **Research Methods**

#### **Participant**

The trial is expected to last for 1 year, with a research period ending on December 31, 2024. It aims to recruit 600 participants, including 150 healthy volunteers to be solicited through advertisements. Additionally, 150 participants with Laryngopharyngeal Reflux (LPR) will be recruited from the Gastroenterology Outpatient Department, along with 150 participants with Functional Dyspepsia (FD) and 150 participants with Irritable Bowel Syndrome (IBS). The inclusion and exclusion criteria for participants are as follows:

### **Inclusion Criteria for Participants:**

#### **Inclusion criteria for healthy subjects:**

- 1. Aged between 18 and 70 years old, clear consciousness, and willing to sign the informed consent form for the study.
- 2. Without any gastrointestinal symptoms or the use of gastrointestinal medications.

#### Inclusion criteria for Laryngopharyngeal reflux disease subject:

- 1. Aged between 18 and 70 years old, clear consciousness, and willing to sign the informed consent form for the study.
- 2. The definition of Laryngopharyngeal Reflux (LPR) is characterized by the presence of symptoms lasting for more than three months, including hoarseness, a sensation of a lump in the throat, chronic cough, and frequent throat clearing. These symptoms occur at least once a week. Diagnosis is confirmed through a standardized LPR assessment questionnaire (Reflux Symptom Index RSI), which consists of nine reflux-related symptoms. Each symptom is rated on a severity scale from 0 (asymptomatic) to 5 (most severe). If the total score exceeds 13 points, the patient meets the criteria for Laryngopharyngeal Reflux.

#### **Inclusion criteria for Functional dyspepsia subject**:

- 1. Aged between 18 and 70 years old, clear consciousness, and willing to sign the informed consent form for the study.
- 2. Those who meet the FD definition Functional dyspepsia is characterized by chronic (occurring at least once a week, lasting for a minimum of three months, with the first symptoms manifesting at least six months ago) upper gastrointestinal symptoms (any of the following): postprandial bloating, a tendency to feel full easily, upper abdominal pain or a burning sensation, without symptoms of gastrointestinal bleeding or significant weight loss, and with no abnormalities found upon upper gastrointestinal endoscopic examination.

#### Inclusion criteria for Irritable bowel syndrome subject:

- 1. Aged between 18 and 70 years old, clear consciousness, and willing to sign the informed consent form for the study.
- 2. Those who meet the definition of IBS. Irritable bowel syndrome (IBS) is a chronic condition characterized by lower gastrointestinal symptoms occurring at least once a week and lasting for a minimum of three months. These symptoms include abdominal pain accompanied by either diarrhea or constipation, without any signs of gastrointestinal bleeding or significant weight loss. Individuals with IBS exhibit no abnormalities upon examination through colonoscopy.

# **Exclusion Criteria for Participants:**

- 1. Pregnant or lactating women.
- 2. Infection currently undergoing antibiotic treatment.
- 3. In the past two months, underwent tracheal intubation.
- 4. Those with myocardial hypoxia or who have recently experienced a myocardial infarction.
- 5. Unable to collaborate.

#### **Research Process Diagram**



Finish experiment

# **Research Steps**

The subjects who meet the inclusion criteria of this study will undergo an initial assessment of heart rate variability and psychosomatic symptoms after enrollment. Subsequently, a two-week

experiment will be conducted, during which the subjects will receive one session of diaphragmatic breathing training by the researchers. After the guided training, the subjects will undergo another assessment of heart rate variability. In the first week, participants will engage in self-practice of the instructed content twice daily, each session lasting 5 minutes, and will record a weekly diaphragmatic breathing diary.

After the first week, subjects will undergo another assessment of heart rate variability and psychosomatic symptoms. In the second week, participants will continue daily self-practice with two sessions of instructed content, each lasting 5 minutes, and will maintain a diaphragmatic breathing diary. Following the second week, subjects will undergo a final assessment of heart rate variability and psychosomatic symptoms, completing the experiment.

Researchers recommend spending approximately 15 minutes on diaphragmatic breathing training, 15 minutes on measuring heart rate variability, and approximately 20 minutes for questionnaire completion. The measurement of heart rate variability utilizes a non-invasive device called "LEADTEK" portable electrocardiogram recorder (Ministry of Health and Welfare Medical Device Manufacturing License No. 006972). If participants have any questions or concerns during the abdominal breathing training process, they are encouraged to contact the researchers.

#### **Diaphragmatic Breathing (It takes about 15 minutes)**

- 1. Sit in a comfortable place and close your eyes.
- **2.** Place one hand on the chest and the other hand on the abdomen to practice diaphragmatic breathing: During diaphragmatic breathing exercises, the hand on the abdomen will rise with inhalation and fall with exhalation, while the hand on the chest remains stationary.
- **3.** Inhale through the nose for about 4 seconds, feeling the expansion of the abdomen. (Upon the first inhalation, there may be a slight sense of tension.)
- **4.** Hold your breath for 2 seconds.
- **5.** Exhale slowly and steadily through the mouth for approximately 6 seconds, keeping the mouth relaxed throughout the process.
- **6.** Repeat this breathing cycle for 5 minutes.

#### **ANS Protocol (It takes about 15 minutes)**

The ANS Protocol is a standardized and validated method used to assess the autonomic nervous system's (ANS) responses to baseline conditions and stress stimuli. It consists of three stages: a resting phase (5 minutes), a mental arithmetic test under stress conditions (3 minutes), and a recovery period (5 minutes) during which heart rate variability (HRV) is measured. The mental arithmetic test involves subjects performing continuous subtraction of 7 from a randomly generated four-digit number using mental calculation only. If an error occurs, the process is restarted, and the entire procedure lasts for 3 minutes.<sup>36</sup>

#### ANS Detection Steps:

- 1. Confirm that the status indicator light is in a measurable state (LED color: green), and then attach the electrode patches. •
- 2. R (Red dot): Please paste on the inner side of the right wrist.
- 3. L (Yellow dot): Please paste on the inner side of the left wrist.
- 4. F (Green Marking): Please paste on the inside of the left wrist.
- 5. Press the measurement button on the device to initiate the measurement.
- 6. Before the formal commencement of measurements, the device will conduct a preliminary signal quality check. Participants are advised to remain still and refrain from engaging in conversation during this process.
- 7. The measurement officially begins at 7: Please instruct the subjects to remain still and refrain from talking, waiting quietly for 3 to 5 minutes until the measurement is completed. •
- 8. Measurement Completed: Display Measurement Results.

The HRV indicators for assessing the ANS are as follows: 21

#### 1. Time Domain Indicators

♦ The square root of the mean of the sum of the squares of the Successive differences (RMSSD): Assessing Parasympathetic Nervous System Activity

#### 2. Frequency Domain Indicators

- ♦ Low frequency power (LF): Assessing Sympathetic Nervous System Activity
- ♦ High frequency power (HF): Assessing Parasympathetic Nervous System Activity
- ♦ Low-frequency/High-frequency Power Ratio (LF/HF ratio) : Assessing the balance of the sympathetic and parasympathetic nervous systems.

#### **Questionnaire Evaluation Tool (It takes about 20 minutes)**

Disease Questionnaire Assessment:

- Gastroesophageal Reflux Disease Questionnaire (GERDQ)<sup>37</sup> The questionnaire score exceeding 12 points indicates a high likelihood of having GERD.
- Reflux Symptom Index (RSI) <sup>38</sup> The nine reflux-related symptoms are graded on a severity scale from 0 (no symptoms) to 5 (most severe), and a total score exceeding 13 indicates a higher probability of suffering from laryngopharyngeal reflux.
- Functional Dyspepsia (FD)<sup>39</sup> The subjective assessment revolves around symptoms and quality of life, primarily including postprandial fullness, early satiety, and upper abdominal bloating as digestive discomfort symptoms. Each item is scored from 0 to 6 points, with 0 points indicating no symptoms and 6 points indicating extremely severe symptoms. The total score ranges from 0 to 52 points, with higher scores indicating more severe symptoms.
- Irritable Bowel Syndrome (IBS)<sup>39</sup> Diagnostic criteria reference Rome IV, The main symptoms began at least 6 months ago, with recurrent abdominal pain occurring at least once a week on average in the past three months. Additionally, at least two of the following symptoms are present: abdominal pain related to bowel movements, changes in bowel frequency, and alterations in the appearance of stool.
- Gastrointestinal Symptom Rating Scale (GSRS)<sup>40</sup> Applicable to the general population with gastrointestinal symptoms for measurement and evaluation of treatment effectiveness, using a Likert 4-point scoring system. Positive scoring is employed, where higher scores indicate greater severity of symptoms, and lower scores represent higher levels of health.

Physical and Mental Stress Questionnaire Assessment:

- Pittsburgh Sleep Quality Index (PSQI) 41 is not only suitable for evaluating sleep quality of patients with sleep disorders and mental disorders, but also suitable for the evaluation of sleep quality of ordinary people. 18 items are composed of 7 components, each component is scored on a scale of 0-3, and the total score ranges from 0-21 points. The higher the score, the worse the sleep quality.
- Taiwanese Depression Scale (TDQ) 42 includes three parts: emotion, cognition and body, with a total of 18 questions, and the scale is scored on a four-point scale. Each question is scored on a scale from 0 to 3, and the total score ranges from 0 to 54 points. Those with a score greater than 18 indicate depressive symptoms.
- State-Trait Anxiety. Inventory (STAI) 43 includes two subscales, the Situational and Trait Anxiety Scale, with a minimum score of 20 and a maximum score of 80, with higher scores representing anxiety symptoms.
- The Perceived Stress Scale (PSS-10) 44 is to evaluate the degree of stress in personal life situations, and the higher the score, the greater the stress.
- Esophageal Hypervigilance and Anxiety Scale (EHAS) 41 Esophageal hypervigilance and anxiety can cause symptoms in patients with chronic esophageal diseases, including gastroesophageal reflux, esophageal atlasia and functional esophageal diseases. The questionnaire contains 15 items and can be divided into two main categories. Section: Symptoms of Esophageal Hypervigilance and Symptoms of Esophageal Anxiety. This questionnaire can not only assess the sensory system symptoms of any esophagus-related diseases, but also assist in the diagnosis of functional esophageal diseases.
- Laryngeal Hypervigilance and Anxiety Scale (LHAS) 41 Throat hypervigilance and anxiety
  can trigger symptoms in patients with chronic esophageal disease. The questionnaire contains
  15 items and can be divided into two main parts: throat hypervigilance symptoms and throat
  anxiety symptoms. This questionnaire can not only assess the sensory system symptoms of
  any esophagus-related diseases, but also assist in the diagnosis of functional esophageal
  diseases.
- Visceral Sensitivity Index (VSI) 45 measures anxiety specific to the gastrointestinal tract. It includes 15 items, with a minimum score of 0 and a maximum of 5 points for each item, and a minimum score of 0 and a maximum score of 75 points for the total score.

#### **Statistical Analysis**

If a continuous variable follows a normal distribution, it is represented by the mean and standard deviation; if it does not follow a normal distribution, it is represented by the median and interquartile range. The treatment effectiveness is presented as the improvement percentage based on the pre- and post-treatment sleep habit questionnaire, depression questionnaire, anxiety questionnaire, stress questionnaire, digestive symptom questionnaire, and irritable bowel syndrome questionnaire. The efficacy of diaphragmatic breathing was assessed using a Chi-squared test to compare percentages. A P-value less than 0.05 was considered statistically significant. The statistical analysis software used is SPSS 19 (SPSS, Inc, Chicago, IL, USA).

# The clinical significance and originality of this study

This study will be the first to extensively apply diaphragmatic breathing to the management of functional gastrointestinal disorders (FGIDs). In addition to assessing gastrointestinal symptoms, it will also evaluate physical and mental symptoms, sleep quality, stress indicators, and visceral sensitivity. Further understanding of autonomic nervous system changes through heart rate variability (HRV). This study aims to investigate the efficacy and mechanism of non-invasive, non-pharmacological diaphragmatic breathing on patients with disorders of the gut-brain axis (DGBI).

# I. Expected deliverables and specific outcomes of the planned tasks

- 1. Please list the work items expected to be completed within the implementation period.
- 2. Anticipated contributions to academic research and other applications.
- 3. For participating staff, the training expected to be available.

#### 1. Expected tasks to be completed

This study expects that diaphragmatic breathing may potentially improve the psychosomatic symptoms of Disorders of Gut-Brain Interaction (DGBI), and it may be achieved by altering autonomic nervous system regulation.

# 2. Expected contributions to academic research, national development, and other applications

The results of this study will provide empirical evidence for the use of diaphragmatic breathing in the treatment of disorders of the gut-brain axis (DGBI). In the future, we hope to participate in the evaluation of the National Healthcare Quality Awards by the Taiwan Medical Association to help a large number of DGBI patients.

#### 3. Expected training for participating staff

Participants will receive not only general research training, such as experimental design and execution, result analysis and statistics, data visualization, oral presentations, paper writing, and manuscript submission process, but also have the opportunity to gain exposure to various experimental techniques and skills due to the diversity of their tasks.

#### J. References

1. Margolis KG, Cryan JF, Mayer EA. The Microbiota-Gut-Brain Axis: From Motility to Mood. Gastroenterology 2021;160:1486-1501.

- 2. Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology 2016;150:1257-61.
- 3. Wong MW, Hsiao SH, Wang JH, et al. Esophageal Hypervigilance and Visceral Anxiety Contribute to Symptom Severity of Laryngopharyngeal Reflux. Am J Gastroenterol 2023;118:786-793.
- 4. Drossman DA, Tack J, Ford AC, et al. Neuromodulators for Functional Gastrointestinal Disorders (Disorders of Gut-Brain Interaction): A Rome Foundation Working Team Report. Gastroenterology 2018;154:1140-1171 e1.
- 5. Duan H, Cai X, Luan Y, et al. Regulation of the Autonomic Nervous System on Intestine. Front Physiol 2021;12:700129.
- 6. Phillips RJ, Powley TL. Innervation of the gastrointestinal tract: patterns of aging. Auton Neurosci 2007;136:1-19.
- 7. Agusti A, Garcia-Pardo MP, Lopez-Almela I, et al. Interplay Between the Gut-Brain Axis, Obesity and Cognitive Function. Front Neurosci 2018;12:155.
- 8. Callaghan B, Furness JB, Pustovit RV. Neural pathways for colorectal control, relevance to spinal cord injury and treatment: a narrative review. Spinal Cord 2018;56:199-205.
- 9. Rao M, Gershon MD. The bowel and beyond: the enteric nervous system in neurological disorders. Nat Rev Gastroenterol Hepatol 2016;13:517-28.
- 10. Carabotti M, Scirocco A, Maselli MA, et al. The gut-brain axis: interactions between enteric microbiota, central and enteric nervous systems. Ann Gastroenterol 2015;28:203-209.
- 11. Browning KN, Travagli RA. Central control of gastrointestinal motility. Curr Opin Endocrinol Diabetes Obes 2019;26:11-16.
- 12. Browning KN, Travagli RA. Central nervous system control of gastrointestinal motility and secretion and modulation of gastrointestinal functions. Compr Physiol 2014;4:1339-68.
- 13. Ali MK, Saha S, Milkova N, et al. Modulation of the autonomic nervous system by one session of spinal low-level laser therapy in patients with chronic colonic motility dysfunction. Front Neurosci 2022;16:882602.
- 14. Ali MK, Chen JDZ. Roles of Heart Rate Variability in Assessing Autonomic Nervous System in Functional Gastrointestinal Disorders: A Systematic Review. Diagnostics (Basel) 2023;13.
- 15. Yuan Y, Ali MK, Mathewson KJ, et al. Associations Between Colonic Motor Patterns and Autonomic Nervous System Activity Assessed by High-Resolution Manometry and Concurrent Heart Rate Variability. Front Neurosci 2019;13:1447.
- 16. Ali MK, Liu L, Chen JH, et al. Optimizing Autonomic Function Analysis via Heart Rate Variability Associated With Motor Activity of the Human Colon. Front Physiol 2021;12:619722.
- 17. Chen J. Neuromodulation and Neurostimulation for the Treatment of Functional Gastrointestinal Disorders. Gastroenterol Hepatol (N Y) 2022;18:47-49.
- 18. Yu Y, Wei R, Liu Z, et al. Ameliorating Effects of Transcutaneous Electrical Acustimulation Combined With Deep Breathing Training on Refractory Gastroesophageal Reflux Disease Mediated via the Autonomic Pathway. Neuromodulation 2019;22:751-757.
- 19. Huang WJ, Shu CH, Chou KT, et al. Evaluating the autonomic nervous system in patients with laryngopharyngeal reflux. Otolaryngol Head Neck Surg 2013;148:997-1002.
- 20. Ouyang H, Yin J, Wang Z, et al. Electroacupuncture accelerates gastric emptying in association with changes in vagal activity. Am J Physiol Gastrointest Liver Physiol 2002;282:G390-6.
- 21. Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health 2017;5:258.
- 22. Shaffer F, McCraty R, Zerr CL. A healthy heart is not a metronome: an integrative review of the heart's anatomy and heart rate variability. Front Psychol 2014;5:1040.
- 23. Ciccone AB, Siedlik JA, Wecht JM, et al. Reminder: RMSSD and SD1 are identical heart rate

- variability metrics. Muscle Nerve 2017;56:674-678.
- 24. Bigger JT, Jr., Albrecht P, Steinman RC, et al. Comparison of time- and frequency domain-based measures of cardiac parasympathetic activity in Holter recordings after myocardial infarction. Am J Cardiol 1989;64:536-8.
- 25. DeGiorgio CM, Miller P, Meymandi S, et al. RMSSD, a measure of vagus-mediated heart rate variability, is associated with risk factors for SUDEP: the SUDEP-7 Inventory. Epilepsy Behav 2010;19:78-81.
- 26. Umetani K, Singer DH, McCraty R, et al. Twenty-four hour time domain heart rate variability and heart rate: relations to age and gender over nine decades. J Am Coll Cardiol 1998;31:593-601.
- 27. Otzenberger H, Gronfier C, Simon C, et al. Dynamic heart rate variability: a tool for exploring sympathovagal balance continuously during sleep in men. Am J Physiol 1998;275:H946-50.
- 28. Karemaker JM. Counterpoint: respiratory sinus arrhythmia is due to the baroreflex mechanism. J Appl Physiol (1985) 2009;106:1742-3; discussion 1744.
- 29. Kocjan J, Adamek M, Gzik-Zroska B, et al. Network of breathing. Multifunctional role of the diaphragm: a review. Adv Respir Med 2017;85:224-232.
- 30. Stauss HM. Heart rate variability. Am J Physiol Regul Integr Comp Physiol 2003;285:R927-31
- 31. Ambrosino N, Paggiaro PL, Macchi M, et al. A study of short-term effect of rehabilitative therapy in chronic obstructive pulmonary disease. Respiration 1981;41:40-4.
- 32. Montano N, Cogliati C, Porta A, et al. Central vagotonic effects of atropine modulate spectral oscillations of sympathetic nerve activity. Circulation 1998;98:1394-9.
- 33. Bernardi L, Gabutti A, Porta C, et al. Slow breathing reduces chemoreflex response to hypoxia and hypercapnia, and increases baroreflex sensitivity. J Hypertens 2001;19:2221-9.
- 34. Yadlapati R, Gyawali CP, Pandolfino JE, et al. AGA Clinical Practice Update on the Personalized Approach to the Evaluation and Management of GERD: Expert Review. Clin Gastroenterol Hepatol 2022;20:984-994 e1.
- 35. Halland M, Bharucha AE, Crowell MD, et al. Effects of Diaphragmatic Breathing on the Pathophysiology and Treatment of Upright Gastroesophageal Reflux: A Randomized Controlled Trial. Am J Gastroenterol 2021;116:86-94.
- 36. Naliboff BD, Benton D, Solomon GF, et al. Immunological changes in young and old adults during brief laboratory stress. Psychosom Med 1991;53:121-32.
- 37. Jones R, Junghard O, Dent J, et al. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther 2009;30:1030-8.
- 38. Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice 2002;16:274-7.
- 39. Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology 2016.
- 40. Revicki DA, Wood M, Wiklund I, et al. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res 1998;7:75-83.
- 41. Taft TH, Triggs JR, Carlson DA, et al. Validation of the oesophageal hypervigilance and anxiety scale for chronic oesophageal disease. Aliment Pharmacol Ther 2018;47:1270-1277.
- 42. Lee Y, Yang MJ, Lai TJ, et al. Development of the Taiwanese Depression Questionnaire. Chang Gung Med J 2000;23:688-94.
- 43. Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken) 2011;63 Suppl 11:S467-72.
- 44. Taylor JM. Psychometric analysis of the Ten-Item Perceived Stress Scale. Psychol Assess 2015;27:90-101.
- 45. Labus JS, Bolus R, Chang L, et al. The Visceral Sensitivity Index: development and validation of a gastrointestinal symptom-specific anxiety scale. Aliment Pharmacol Ther 2004;20:89-97.